CLINICAL TRIAL: NCT07267572
Title: Randomized, Comparative Study to Evaluate the Added Value of Logotherapy in the Psychological Support of Patients With Primary Breast Cancer
Brief Title: Evaluation of the Added Value of Logotherapy in the Psychological Support of Patients With Primary Breast Cancer
Acronym: AELO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Elsan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AELO; 2024-A02252-45 (Other: ANSM)
Record Dates: First submitted 2025-11-25; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer
Keywords: logotherapy; support; breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Logotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Support within the framework of the "announcement procedure" with logotherapy (Experimental)
  Interventions: Other: Support to the patient including logotherapy
- Support within the framework of the "announcement procedure" without logotherapy (Active Comparator)
  Interventions: Other: Support to the patient without logotherapy

INTERVENTIONS:
Other: Support to the patient including logotherapy — Logotherapy consists of four individual sessions conducted by a nurse who is specialized and certified in logotherapy, at a rate of one session every two weeks, lasting approximately 60 minutes.
  Arms: Support within the framework of the "announcement procedure" with logotherapy
Other: Support to the patient without logotherapy — Supportive care offered as part of the patient notification process following the diagnosis of breast cancer.
  Arms: Support within the framework of the "announcement procedure" without logotherapy

SUMMARY:
The diagnosis of breast cancer in a woman can cause major psychological trauma with many destructive effects in all areas of life.

Dealing with this profound distress is often difficult, sometimes poorly defined between different professionals (psychiatrists, psychologists, psychotherapists, proponents of alternative therapies), leading to highly variable and difficult-to-measure results.

Since the first French cancer plan (2003/2007), facilities offering cancer care have been legally required to have a notification and support system in place. This consists of offering patients a range of supportive care throughout their cancer treatment (psychotherapy, physical activities, dietetics, pain management, etc.).

In recent years, logotherapy has been offered as part of psychological care. Logotherapy is a form of psychotherapy based on meaning, which has been offered for many years and aims to help patients create or discover meaning in their lives. Meaning serves as motivation to continue living despite illness by placing this ordeal in the context of existence.

Suffering can thus be transformed into opportunity. The use of logotherapy gives the suffering person the ability to take an active part in their treatment and helps them to mobilize their personal resources to keep the disease at bay, stabilize it, or cure it.

Several studies conducted on women with breast or gynecological cancer have shown that logotherapy can reduce the symptoms of traumatic stress and increase their ability to find meaning in their lives. However, these studies have certain limitations because they are not randomized.

In order to evaluate the short- and medium-term benefits of logotherapy in patients diagnosed with primary breast cancer, we propose a prospective, comparative, randomized study.

ELIGIBILITY:
Inclusion Criteria:

Female patient:

* With a first diagnosis of histologically proven breast cancer,
* Affiliated to a health insurance scheme,
* Having been informed and having given her free and informed consent prior to any procedure specific to the study.

Exclusion Criteria:

Female patient:

* Unable to understand the study and to answer to the questionnaires
* With an indication for neoadjuvant chemotherapy
* Undergoing antidepressant treatment at the time of diagnosis
* Presenting with alcohol or drug addiction at the time of diagnosis
* Protected: adult under guardianship, curatorship, or other legal protection, deprived of liberty by judicial or administrative decision.
* Pregnant, breastfeeding, or in labor.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Anxiety | 10 weeks
  Anxiety score of the Hospital Anxiety and Depression Scale (HADS) score. The HADS is a validated self-administered questionnaire consisting of 14 items allowing patients to assess their mood over the past week. It is composed of two parts (anxiety and depression) The result ranges from 0 to 21.
Depression | 10 weeks
  Depression score of the HADS. This score will be analysed on a second step (two-step hierarchical sequential analysis) only if a significative difference is observable on the first step (anxiety).

SECONDARY OUTCOMES:
Anxiety and depression | Baseline, 10 weeks, 6 months and 9 months
  HADS score (anxiety and depression).
Perceived stress | Baseline, 10 weeks, 6 months and 9 months
  Perceived Stress Scale (PSS) score. It is a validated self-administered questionnaire, comprising 10 questions assessing a patient's individual stress level. The result is expressed in a score between 0 (no perceived stress) and 40 (high perceived stress)
Quality of life assessment | Baseline, 10 weeks, 6 months and 9 months
  EORTC QJQ-C30. It is a general self-administered questionnaire comprising 30 questions to assess the quality of life of cancer patients participating in clinical trials. The result is expressed in a score between 0 and 100.
Consultations of psychotherapists | Over 9 months
  Number of consultations with a specialist in psychotherapy in relation to breast cancer management.
Anxyolitic treatments consumption | 10 weeks, 6 months and 9 months
  Number of anxyolitic treatments (type, dose and indication)
Anti-depressant treatments consumption | 10 weeks, 6 months and 9 months
  Number of anti-depressant treatments (type, dose and indication)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique du Fief de Grimoire, Poitiers, France

IPD SHARING:
Plan to Share IPD: No